CLINICAL TRIAL: NCT01623934
Title: Role of Adipokines in Glucose Regulation During Pregnancy and in Fetal Development
Acronym: GEN3G
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); American Diabetes Association (Other); Diabetes Québec (Other)
Responsible Party: Principal Investigator, Marie-France Hivert, Md, MMSc, Université de Sherbrooke
Other Study IDs: GEN3G
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Gestational Diabetes; Insulin Resistance; Obesity Prevention
Keywords: Gestational diabetes; Adiponectin; Leptin; Single Nucleotides Polymorphisms; Insulin resistance; obesity
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal and child plasma, whole cord blood, serum/plasma cord blood, maternal and child white cells, placenta, maternal and child urine, child saliva, maternal and child stool, child hair
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phase 1: Pregnant women
- Phase 2: Mother-offspring dyad

SUMMARY:
This study includes 2 phases. During phase 1, pregnant women are followed over the course of pregnancy. The phase 2 is a follow-up of the mother-child dyad at 3, 5 and 10-12 year after delivery.

The purpose of this phase 1 is to :

* assess the contribution and interactions of adipokines in the development of insulin resistance during pregnancy and gestational diabetes;
* assess levels of maternal adipokines as determinants of development and fetal growth;
* determine the genetic variations that influence levels of adipokines and glucose regulation during pregnancy and in newborns.

The purpose of this phase 2 is to:

* identify DNA methylation variations at birth that are predictive of childhood overweight/obesity.
* identify maternal characteristics associated with DNA methylation variations predictive of childhood overweight/obesity.
* establish whether the loci predictive of childhood overweight/obesity at birth are still differentially methylated at 5 years of age (samples collected at 5 years of age).
* identify DNA methylation variations at birth that are predictive of childhood neurodevelopment problems at 3, 5 and 10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 yrs
* gestational age between 6 and 13 weeks from last menstrual period
* no recognized diabetes or drugs interfering with glucose metabolism
* alcohol < 2 drinks/day
* not involved in regular high intensity physical activity
* otherwise good health status

Exclusion Criteria:

* twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1: Pregnant women when they come for their first prenatal visit at the Clinique de Prélèvements et de Recherche en Grossesse.
  Phase 2: mothers and their child
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2010-01; Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of gestational diabetes mellitus | 24-28 weeks of gestation
  75g oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Hivert, MD, MSc, Principal Investigator — Harvard Medical School, Harvard Prilgrim Health Care Institute
Locations (1):
- Centre de recherche du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Guillemette L, Allard C, Lacroix M, Patenaude J, Battista MC, Doyon M, Moreau J, Menard J, Bouchard L, Ardilouze JL, Perron P, Hivert MF. Genetics of Glucose regulation in Gestation and Growth (Gen3G): a prospective prebirth cohort of mother-child pairs in Sherbrooke, Canada. BMJ Open. 2016 Feb 3;6(2):e010031. doi: 10.1136/bmjopen-2015-010031. PMID 26842272